CLINICAL TRIAL: NCT01590576
Title: Population-based Estimates of Medical Comorbidities in Women With Lower Urinary Tract Symptoms or Pelvic Organ Prolapse
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Sheng-Mou Hsiao, Chief, Department of Obstetrics & Gynecology, Far Eastern Memorial Hospital
Other Study IDs: 101019-E
Record Dates: First submitted 2012-05-01; First posted 2012-05-03 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-02

CONDITIONS: Lower Urinary Tract Symptoms; Pelvic Organ Prolapse
Keywords: women
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Pelvic Organ Prolapse

STUDY DESIGN:
Time Perspective: Retrospective

GROUPS / COHORTS (1):
- lower urinary tract symptoms and pelvic organ prolapse

SUMMARY:
The purpose of this study is to investigate the comorbidities of lower urinary tract symptoms or pelvic organ prolapse in a nationwide population-based data in Taiwan during the study period of 2001-2010, a total of 10 years.

ELIGIBILITY:
Inclusion Criteria:

* all cases with lower urinary tract symptoms

Ages: 20 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with low urinary tract symptoms
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Actual)
Dates: Start 2014-11; Primary Completion 2016-01 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Far-Eastern Memorial Hospital, Banqiao District, New Taipei, Taiwan